CLINICAL TRIAL: NCT00094458
Title: Multicenter, Randomized, Double-Blind, Active Controlled Trial Comparing REMICADE� (Infliximab) and REMICADE Plus Azathioprine to Azathioprine in the Treatment of Patients With Crohn's Disease Naive to Both Immunomodulators and Biologic Therapy
Brief Title: Trial Comparing Infliximab and Infliximab and Azathioprine in the Treatment of Patients With Crohn's Disease na�ve to Both Immunomodulators and Biologic Therapy (Study of Biologic and Immunomodulator Naive Patients in Chrohn's Disease: SONIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor Ortho Biotech Services, L.L.C. (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR004804; C0168T67
Record Dates: First submitted 2004-10-19; First posted 2004-10-20 (Estimated); Results first posted 2009-06-23 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; infliximab; azathioprine; Remicade; SONIC
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab; Azathioprine; Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 003 (Experimental): infliximab (IFX) infusion; azathioprine (AZA) caps AZA daily 2.5 mg/kg/day and IFX infusions 5 mg/kg at weeks 0, 2, 6, 14, and 22
  Interventions: Other: infliximab (IFX) infusion; azathioprine (AZA) caps
- 001 (Experimental): infliximab (IFX) placebo infusion; azathioprine (AZA) caps AZA daily 2.5 mg/kg/day and placebo IFX infusions at weeks 0, 2, 6, 14, and 22
  Interventions: Drug: infliximab (IFX) placebo infusion; azathioprine (AZA) caps
- 002 (Experimental): infliximab infusion; AZA placebo caps Infliximab 5 mg/kg at weeks 0, 2, 6, 14, and 22 and placebo AZA capsules
  Interventions: Biological: infliximab infusion; AZA placebo caps

INTERVENTIONS:
Biological: infliximab infusion; AZA placebo caps — Infliximab 5 mg/kg at weeks 0, 2, 6, 14, and 22 and placebo AZA capsules
  Arms: 002
Other: infliximab (IFX) infusion; azathioprine (AZA) caps — AZA daily 2.5 mg/kg/day and IFX infusions 5 mg/kg at weeks 0, 2, 6, 14, and 22
  Arms: 003
Drug: infliximab (IFX) placebo infusion; azathioprine (AZA) caps — AZA daily 2.5 mg/kg/day and placebo IFX infusions at weeks 0, 2, 6, 14, and 22
  Arms: 001

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of three different treatments for patients with Crohns disease who have not responded to previous treatment with a group of drugs commonly used to treat Crohn's Disease (5-ASA) and corticosteroids. Patients will receive either infliximab (a drug used to treat autoimmune diseases) or azathioprine (an immunosuppressant or drug used to suppress the immune system) or a combination of both for up to 34 weeks. This research study will involve approximately 500 patients. The main study involves up to 34 weeks (approximately 8 months). A study extension of an additional 20 weeks (approximately 5 months) is optional for patients who successfully complete the main study. A country-specific study extension of open label infliximab treatment for an additional 1 year is optional for patients who successfully complete the main study extension.

DETAILED DESCRIPTION:
Crohns disease is characterized by inflammation (the changes that happen when tissues in the body are injured) and ulceration (open sores) of the intestines. Crohns disease is treated with medications that decrease inflammation, and reduce diarrhea, abdominal pain and other symptoms of Crohns disease. In addition, Crohns disease can be treated with medications that suppress the immune system (the body system involved in inflammation and infections) or with surgery. This study will investigate the effectiveness of infliximab and azathioprine in the treatment of patients with moderate-to-severe Crohns disease. Infliximab is currently approved by the FDA for the treatment of both Crohns disease and rheumatoid arthritis. Azathioprine, which is an investigational drug, has not been approved by the FDA for the treatment of Crohns disease, but it is a well-established therapy that has been used for many years to treat Crohns disease. This study seeks to determine whether infliximab, azathioprine, or the combination of both drugs would be the most appropriate treatment for Crohns disease patients who have not responded well to certain drugs called 5-ASA drugs (e.g. Asacol, Pentasa, sulfasalazine) and/or require frequent treatment with corticosteroids. This research study will involve approximately 500 patients. Patients may participate in the main study for up to 34 weeks (approximately 8 months). During the main study, patients will be asked to visit the study center for 10 visits. If patients enroll into the extension of the study, the total time for participation may be up to 54 weeks (approximately 13 months). Patients enrolled in the Study Extension will be asked to visit the study center for an additional 5 visits. A country-specific (EU and Israel only), prospective, multi-center, open-label extension of the study will further evaluate the long-term safety and efficacy of scheduled maintenance therapy with infliximab in patients with Crohns Disease. Patients who have completed treatment through Week 50 in the SONIC main study and who, in the opinion of the investigator, would benefit from infliximab treatment may enter the open-label extension. Patients will be randomly assigned to one of three treatment groups (either infliximab plus placebo capsules, infliximab plus azathioprine, or azathioprine plus placebo infusions - there is no possibility of being assigned to placebo only in this trial - patients will receive one or both of these medications) at the beginning of the study. Oral medication will be taken daily. There are 5 infusion (which will be either infliximab or placebo) visits during the main study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohns Disease for at least 6 weeks
* Moderate to severe disease activity (CDAI >= 220 and <=450)
* No history of azathioprine, 6-MP (6 Mercaptopurine), or biologic treatments
* Are either: Corticosteriod-dependent, OR considered for a 2nd (or greater) course of corticosteriod, OR 5-ASA failures, Or Budesonide failures

Exclusion Criteria:

* History of abdominal surgery within the last 6 months
* Have an ostomy or stoma [An operation to create an opening from an area inside the body to the outside]
* Are pregnant, nursing, or planning pregnancy (both men and women)
* Serious simultaneous illness that could interfere with study participation
* Use of any investigational drug within 30 days
* Have a concomitant diagnosis or any history of congestive heart failure
* Weigh more than 140 kilograms (or 310 pounds)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2005-03; Primary Completion 2008-04 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor Ortho Biotech Services, L.L.C. Clinical Trial, Study Director — Centocor Ortho Biotech Services, L.L.C.
Locations (115):
- United States (51):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Orange, California
  - Roseville, California
  - San Diego, California
  - San Luis Obispo, California
  - Golden, Colorado
  - Littleton, Colorado
  - Hartford, Connecticut
  - Gainesville, Florida
  - Jacksonville, Florida
  - North Miami Beach, Florida
  - Winter Park, Florida
  - Austell, Georgia
  - Decatur, Georgia
  - Savannah, Georgia
  - Peoria, Illinois
  - Clive, Iowa
  - Overland Park, Kansas
  - Topeka, Kansas
  - Baton Rouge, Louisiana
  - Metairie, Louisiana
  - Troy, Michigan
  - Plymouth, Minnesota
  - Rochester, Minnesota
  - Ocean Springs, Mississippi
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Urbana, Missouri
  - Lincoln, Nebraska
  - Egg Harbor, New Jersey
  - Great Neck, New York
  - New Hyde Park, New York
  - New York, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Bend, Oregon
  - Portland, Oregon
  - Hatfield, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Columbia, South Carolina
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Bellevue, Washington
  - Spokane, Washington
  - Tacoma, Washington
- Austria (2):
  - Hall in Tirol
  - Vienna
- Belgium (5):
  - Bonheiden
  - Brussels
  - Leuven
  - Liège
  - Roeselare
- Canada (3):
  - Montreal, Ontario
  - Toronto, Ontario
  - Québec, Quebec
- Denmark (3):
  - Aalborg
  - Aarhus C
  - Helsinge
- France (8):
  - Amiens
  - Bordeaux
  - Caen
  - Grenoble
  - Lille
  - Nancy
  - Paris
  - Toulouse
- Germany (11):
  - Berlin
  - Frankfurt am Main
  - Hamburg
  - Hanover
  - Herne
  - Kiel
  - Magdeburg
  - Mainz
  - Minden
  - München
  - Münster
- Greece (4):
  - Athens
  - Eksochi
  - Heraklion- Crete
  - Nicea
- Israel (5):
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Tel Aviv
- Netherlands (3):
  - Dordrecht
  - Eindhoven
  - Rotterdam
- Oslo, Norway
- Portugal (2):
  - Amadora
  - Coimbra
- Spain (6):
  - Barcelona
  - Madrid
  - Santander
  - Santiago de Compostela
  - Seville
  - Valencia
- Sweden (4):
  - Linköping
  - Lund
  - Stockhollm
  - Stockholm
- United Kingdom (7):
  - Bristol
  - Cambridge
  - Leeds
  - Livingston
  - London
  - Newcastle upon Tyne
  - Stockport

REFERENCES:
- [Result] Colombel JF, Sandborn WJ, Reinisch W, Mantzaris GJ, Kornbluth A, Rachmilewitz D, Lichtiger S, D'Haens G, Diamond RH, Broussard DL, Tang KL, van der Woude CJ, Rutgeerts P; SONIC Study Group. Infliximab, azathioprine, or combination therapy for Crohn's disease. N Engl J Med. 2010 Apr 15;362(15):1383-95. doi: 10.1056/NEJMoa0904492. PMID 20393175
- [Derived] Dulai PS, Wong ECL, Reinisch W, Narula N. Clinical Decision Support Tool for Infliximab in Crohn's Disease. Clin Gastroenterol Hepatol. 2022 May;20(5):e1192-e1195. doi: 10.1016/j.cgh.2021.06.037. Epub 2021 Jun 30. PMID 34216825
- [Derived] Colombel JF, Adedokun OJ, Gasink C, Gao LL, Cornillie FJ, D'Haens GR, Rutgeerts PJ, Reinisch W, Sandborn WJ, Hanauer SB. Combination Therapy With Infliximab and Azathioprine Improves Infliximab Pharmacokinetic Features and Efficacy: A Post Hoc Analysis. Clin Gastroenterol Hepatol. 2019 Jul;17(8):1525-1532.e1. doi: 10.1016/j.cgh.2018.09.033. Epub 2018 Sep 26. PMID 30267864
- [Derived] Colombel JF, Reinisch W, Mantzaris GJ, Kornbluth A, Rutgeerts P, Tang KL, Oortwijn A, Bevelander GS, Cornillie FJ, Sandborn WJ. Randomised clinical trial: deep remission in biologic and immunomodulator naive patients with Crohn's disease - a SONIC post hoc analysis. Aliment Pharmacol Ther. 2015 Apr;41(8):734-46. doi: 10.1111/apt.13139. Epub 2015 Mar 1. PMID 25728587
- [Derived] Reinisch W, Colombel JF, Sandborn WJ, Mantzaris GJ, Kornbluth A, Adedokun OJ, Miller M, Tang KL, Rutgeerts P, Cornillie F. Factors associated with short- and long-term outcomes of therapy for Crohn's disease. Clin Gastroenterol Hepatol. 2015 Mar;13(3):539-547.e2. doi: 10.1016/j.cgh.2014.09.031. Epub 2014 Sep 19. PMID 25245629
- [Derived] Peyrin-Biroulet L, Reinisch W, Colombel JF, Mantzaris GJ, Kornbluth A, Diamond R, Rutgeerts P, Tang LK, Cornillie FJ, Sandborn WJ. Clinical disease activity, C-reactive protein normalisation and mucosal healing in Crohn's disease in the SONIC trial. Gut. 2014 Jan;63(1):88-95. doi: 10.1136/gutjnl-2013-304984. Epub 2013 Aug 23. PMID 23974954
- [Derived] Ferrante M, Colombel JF, Sandborn WJ, Reinisch W, Mantzaris GJ, Kornbluth A, Rachmilewitz D, Lichtiger S, D'Haens GR, van der Woude CJ, Danese S, Diamond RH, Oortwijn AF, Tang KL, Miller M, Cornillie F, Rutgeerts PJ; International Organization for the Study of Inflammatory Bowel Diseases. Validation of endoscopic activity scores in patients with Crohn's disease based on a post hoc analysis of data from SONIC. Gastroenterology. 2013 Nov;145(5):978-986.e5. doi: 10.1053/j.gastro.2013.08.010. Epub 2013 Aug 14. PMID 23954314

RESULTS

PARTICIPANT FLOW:
Groups:
- Azathioprine + Placebo: Participants received placebo (PBO) infusions and daily Azathioprine (AZA) capsules in main study through Week 30. Participants who completed treatment in the main study and in the opinion of investigator, had benefited from continued treatment were entered in the study extension and received same assigned treatments (which they were receiving in main study) from Week 30 to 46. Those who completed treatment in the study extension may enter in country specific (EU and Israel) OLE.
- Infliximab + Placebo: Participants received infliximab (IFX) infusions 5 mg/kg body weight of participant along with placebo capsules daily in main study through Week 30. Participants who completed treatment in the main study and, in the opinion of investigator, had benefited from continued treatment were entered in the study extension and received same assigned treatments (which they were receiving in main study) from Week 30 to 46. Those who completed treatment in the study extension may enter in country specific (EU and Israel) OLE.
- Infliximab + Azathioprine: Participants received infliximab infusions 5 mg/kg body weight of participant along with daily AZA capsules 2.5 mg/kg body weight of participant in main study through Week 30. Participants who completed treatment in the main study and, in the opinion of investigator, had benefited from continued treatment were entered in the study extension and received same assigned treatments (which they were receiving in main study) from Week 30 to 46. Those who completed treatment in the study extension may enter in country specific (EU and Israel) OLE.
- Azathioprine + Placebo/Infliximab: Participants received daily AZA oral capsules 2.5mg/kg/day and Placebo infusion through Week 50. Infliximab (IFX) infusions 5mg/kg in one year country specific (EU and Israel) open-Label Extension.
- Infliximab + Placebo/Infliximab: Participants received Placebo oral capsules daily and IFX infusions 5mg/kg through Week 50. IFX infusions 5mg/kg in one year country specific (EU and Israel) Open-Label Extension.
- Infliximab + Azathioprine/Infliximab: Participants received daily AZA oral capsules 2.5mg/kg/day and IFX infusions 5mg/kg through Week 50. IFX infusions 5mg/kg in one year country specific (EU and Israel) Open-Label Extension.
Period: Main Study: Through Week 30
Arm/Group | Azathioprine + Placebo | Infliximab + Placebo | Infliximab + Azathioprine | Azathioprine + Placebo/Infliximab | Infliximab + Placebo/Infliximab | Infliximab + Azathioprine/Infliximab
Started | 170 | 169 | 169 | 0 | 0 | 0
Completed | 86 | 111 | 121 | 0 | 0 | 0
Not Completed | 84 | 58 | 48 | 0 | 0 | 0
Not completed — Eligibility criteria not met | 3 | 8 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 5 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 18 | 9 | 7 | 0 | 0 | 0
Not completed — Adverse Event | 38 | 20 | 28 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 19 | 16 | 9 | 0 | 0 | 0
Period: Study Extension: Week 30 Through Week 50
Arm/Group | Azathioprine + Placebo | Infliximab + Placebo | Infliximab + Azathioprine | Azathioprine + Placebo/Infliximab | Infliximab + Placebo/Infliximab | Infliximab + Azathioprine/Infliximab
Started | 75 | 97 | 108 | 0 | 0 | 0
Completed | 67 | 85 | 90 | 0 | 0 | 0
Not Completed | 8 | 12 | 18 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 4 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 9 | 7 | 0 | 0 | 0
Not completed — Other | 1 | 2 | 3 | 0 | 0 | 0
Period: OLE: Open-Label Extension
Arm/Group | Azathioprine + Placebo | Infliximab + Placebo | Infliximab + Azathioprine | Azathioprine + Placebo/Infliximab | Infliximab + Placebo/Infliximab | Infliximab + Azathioprine/Infliximab
Started | 0 | 0 | 0 | 8 | 18 | 17
Completed | 0 | 0 | 0 | 7 | 13 | 13
Not Completed | 0 | 0 | 0 | 1 | 5 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3 | 4
Not completed — Inadequate therapeutic effect | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Patient decision | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azathioprine + Placebo | Infliximab + Placebo | Infliximab + Azathioprine | Total
Number analyzed (Participants) | 170 | 169 | 169 | 508
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (12.92) | 36.6 (13) | 35.9 (11.97) | 36.3 (12.62)
Gender [Count of Participants; unit: Participants]
  Female | 80 | 85 | 81 | 246
  Male | 90 | 84 | 88 | 262
Region of Enrollment [Number; unit: participants]
  AUSTRIA | 8 | 9 | 8 | 25
  BELGIUM | 14 | 17 | 15 | 46
  CANADA | 9 | 7 | 7 | 23
  DENMARK | 5 | 8 | 4 | 17
  FRANCE | 9 | 12 | 18 | 39
  GERMANY | 17 | 8 | 13 | 38
  GREECE | 3 | 3 | 3 | 9
  ISRAEL | 7 | 13 | 12 | 32
  NETHERLANDS | 9 | 9 | 8 | 26
  NORWAY | 0 | 1 | 0 | 1
  PORTUGAL | 0 | 2 | 0 | 2
  SPAIN | 2 | 2 | 2 | 6
  SWEDEN | 0 | 1 | 2 | 3
  UK | 4 | 11 | 7 | 22
  USA | 83 | 66 | 70 | 219

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Corticosteriod-free Clinical Remission
Description: Corticosteroid-free clinical remission is defined as a Crohn's Disease Activity Index (CDAI) less than (<) 150 in participants who have not received any dose of systemic corticosteroids (prednisone or equivalent) for greater than or equal to (>=) 3 weeks and have not received budesonide at a dose > 6 milligram per day (mg/day) for >= 3 weeks. The total CDAI score ranges from 0 - 600. The lower the CDAI score, the better (i.e., 0 is better and 600 is worse).
Time Frame: Week 26
Population: Intention to treat (ITT) population includes all randomized participants in the analysis, according to the treatment group to which they were randomized, regardless of the treatment they actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Azathioprine + Placebo | Infliximab + Placebo | Infliximab + Azathioprine
Number analyzed (Participants) | 170 | 169 | 169
percentage of participants | 30.0 | 44.4 | 56.8
Statistical Analysis 1: Comparison: Azathioprine + Placebo vs Infliximab + Azathioprine; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; The P-Value is from a CMH test stratified by duration of Crohn's disease and corticosteroid treatment at Baseline
Statistical Analysis 2: Comparison: Azathioprine + Placebo vs Infliximab + Placebo; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel; The P-Value is from a CMH test stratified by duration of Crohn's disease and corticosteroid treatment at Baseline
Statistical Analysis 3: Comparison: Infliximab + Placebo vs Infliximab + Azathioprine; Test type: Superiority or Other; p = 0.022, Cochran-Mantel-Haenszel; The P-Value is from a CMH test stratified by duration of Crohn's disease and corticosteroid treatment at Baseline

2. Secondary Outcome: Percentage of Participants With Mucosal Healing
Description: Complete absence of mucosal ulcerations in the colon and terminal ileum as assessed by video endoscopy.
Time Frame: Week 26
Population: Analysis population for mucosal healing was per protocol. All subjects with lesions at Baseline (Week 0) and an Endoscopy at Week 26 were included in the analysis. Here, 'N' [number of participants analyzed] signifies those participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Azathioprine + Placebo | Infliximab + Placebo | Infliximab + Azathioprine
Number analyzed (Participants) | 109 | 93 | 107
percentage of participants | 16.5 | 30.1 | 43.9
Statistical Analysis 1: Comparison: Azathioprine + Placebo vs Infliximab + Azathioprine; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; The P-Value is from a CMH test stratified by duration of Crohn's disease and corticosteroid treatment at Baseline
Statistical Analysis 2: Comparison: Azathioprine + Placebo vs Infliximab + Placebo; Test type: Superiority or Other; p = 0.023, Cochran-Mantel-Haenszel; The P-Value is from a CMH test stratified by duration of Crohn's disease and corticosteroid treatment at Baseline
Statistical Analysis 3: Comparison: Infliximab + Placebo vs Infliximab + Azathioprine; Test type: Superiority or Other; p = 0.055, Cochran-Mantel-Haenszel; The P-Value is from a CMH test stratified by duration of Crohn's disease and corticosteroid treatment at Baseline

3. Secondary Outcome: Percentage of Participants With Corticosteroid-free Clinical Remission (Study Extension)
Description: Corticosteroid-free clinical remission is defined as a Crohn's Disease Activity Index (CDAI) < 150 who have not received any dose of systemic corticosteroids (prednisone or equivalent) for >= 3 weeks and have not received budesonide at a dose > 6 milligram per day (mg/day) for >= 3 weeks. The total CDAI score ranges from 0 - 600. The lower the CDAI score, the better (i.e., 0 is better and 600 is worse).
Time Frame: Week 50
Population: Population analyzed included all randomized participants enrolled in Study Extension.
Measure: Number; unit: percentage of participants
Arm/Group | Azathioprine + Placebo | Infliximab + Placebo | Infliximab + Azathioprine
Number analyzed (Participants) | 75 | 97 | 108
percentage of participants | 54.7 | 60.8 | 72.2

4. Secondary Outcome: Percentage of Participants With Clinical Remission (Main Study)
Description: Clinical remission is defined as a CDAI < 150, compared to baseline (Week 0)
Time Frame: Weeks 2, 6, 10, 18 and 26
Population: Population analyzed included all randomized participants enrolled in the main study.
Measure: Number; unit: percentage of participants
Arm/Group | Azathioprine + Placebo | Infliximab + Placebo | Infliximab + Azathioprine
Number analyzed (Participants) | 170 | 169 | 169
percentage of participants
  Week 2 | 17.6 | 32.5 | 36.7
  Week 6 | 27.6 | 49.1 | 52.1
  Week 10 | 34.1 | 47.3 | 59.8
  Week 18 | 33.5 | 49.7 | 60.4
  Week 26 | 31.8 | 47.9 | 60.4

5. Secondary Outcome: Percentage of Participants With Clinical Remission (Study Extension)
Description: Clinical remission is defined as a CDAI < 150, compared to baseline (Week 0)
Time Frame: Weeks 34, 42 and 50
Population: Population analyzed included all randomized participants enrolled in the Study Extension.
Measure: Number; unit: percentage of participants
Arm/Group | Azathioprine + Placebo | Infliximab + Placebo | Infliximab + Azathioprine
Number analyzed (Participants) | 75 | 97 | 108
percentage of participants
  Week 34 | 61.3 | 66.0 | 69.4
  Week 42 | 58.7 | 72.2 | 73.1
  Week 50 | 54.7 | 66.0 | 74.1

6. Secondary Outcome: Percentage of Participants With Clinical Response Over Time (Main Study)
Description: Clinical response, defined as a >=100-point decrease in CDAI from Baseline.
Time Frame: Weeks 2, 6, 10, 18, 26
Population: Population analyzed included all randomized participants during the Main Study.
Measure: Number; unit: percentage of participants
Arm/Group | Azathioprine + Placebo | Infliximab + Placebo | Infliximab + Azathioprine
Number analyzed (Participants) | 170 | 169 | 169
percentage of participants
  Week 2 | 22.4 | 42.6 | 47.3
  Week 6 | 37.6 | 54.4 | 63.3
  Week 10 | 39.4 | 55.6 | 69.2
  Week 18 | 38.8 | 55.0 | 62.7
  Week 26 | 37.6 | 54.4 | 62.1

7. Secondary Outcome: Percentage of Participants With Clinical Response Over Time (Study Extension)
Description: Clinical response, defined as a >=100-point decrease in CDAI from Baseline.
Time Frame: Weeks 34, 42, 50
Population: Population analyzed included all randomized participants during the Study Extension.
Measure: Number; unit: percentage of participants
Arm/Group | Azathioprine + Placebo | Infliximab + Placebo | Infliximab + Azathioprine
Number analyzed (Participants) | 75 | 97 | 108
percentage of participants
  Week 34 | 66.7 | 76.3 | 76.9
  Week 42 | 65.3 | 74.2 | 77.8
  Week 50 | 62.7 | 72.2 | 78.7

8. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score at Weeks 2, 6, 10, 18 and 26 (Main Study)
Description: Quality of life as measured by the Inflammatory Bowel Disease Questionnaire (IBDQ). The IBDQ is a 32- item questionnaire and the total IBDQ score can range from 32 (very poor) to 224 (perfect).
Time Frame: Baseline and Weeks 2, 6, 10, 18, 26
Population: Population analyzed included all randomized participants enrolled in Main Study with last observation carried forward method to impute missing data. 'n' signifies number of participants who were evaluable at specified time point, for each arm respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azathioprine + Placebo | Infliximab + Placebo | Infliximab + Azathioprine
Number analyzed (Participants) | 170 | 169 | 169
units on a scale
  Week 2 (n= 160, 160, 163) | 20.1 (24.29) | 27.7 (26.08) | 31.4 (29.60)
  Week 6 (n= 162, 161, 165) | 28.3 (31.25) | 34.8 (31.79) | 39.9 (32.90)
  Week 10 (n= 162, 161, 165) | 31.0 (31.66) | 37.8 (35.56) | 42.4 (34.67)
  Week 18 (n= 162, 161, 165) | 30.3 (33.92) | 39.9 (34.17) | 43.7 (34.56)
  Week 26 (n= 162, 161, 165) | 31.4 (35.43) | 39.9 (36.62) | 45.2 (35.76)

9. Secondary Outcome: Average Corticosteroid Use
Description: Average daily dose of systemic corticosteroid concomitant medications(prednisone or equivalent)
Time Frame: Weeks 2, 6, 10, 18 and 26
Population: Population analyzed included all randomized participants taking corticosteroids for Crohn's disease. n' signifies number of participants who were evaluable at specified time point, for each arm respectively.
Measure: Mean (Standard Deviation); unit: milligram per day
Arm/Group | Azathioprine + Placebo | Infliximab + Placebo | Infliximab + Azathioprine
Number analyzed (Participants) | 170 | 169 | 169
milligram per day
  Week 2 (n=48, 50, 49) | 22.92 (12.476) | 21.20 (11.883) | 22.75 (11.923)
  Week 6 (n=53, 52, 51) | 18.56 (11.588) | 17.68 (10.993) | 18.26 (11.635)
  Week 10 (n=56, 56, 52) | 16.19 (11.160) | 15.68 (14.924) | 15.01 (11.087)
  Week 18 (n=59, 57, 56) | 13.49 (10.929) | 13.23 (17.206) | 11.64 (10.904)
  Week 26 (n=60, 60, 58) | 11.57 (10.246) | 10.96 (15.990) | 9.35 (10.052)

ADVERSE EVENTS:
Description: 1 patient in AZA+PBO group(gp),3 in IFX+PBO gp,1 in IFX+AZA gp were randomized but not treated(Excluded from safety analyses).Safety population for IFX+AZA gp included 11 patients assigned to one of monotherapy gps but inadvertently were given at least one dose of both active oral and intravenous therapy(8 patients in AZA+PBO gp,3 in IFX+PBO gp).
Groups:
- W30-Azathioprine + Placebo: Azathioprine (AZA) oral capsules 2.5 mg/kg/day and Placebo (PBO) infusion through Week 30.
- W30-Infliximab + Placebo: Placebo (PBO) oral daily and Infliximab (IFX) infusions 5 mg/kg through Week 30.
- W30-Infliximab + Azathioprine: Azathioprine (AZA) oral daily 2.5 mg/kg/day and Infliximab (IFX) infusions 5mg/kg through Week 30.
- W50-Azathioprine + Placebo: (AZA) oral daily 2.5 mg/kg/day and Placebo (PBO) infusion Week 30 through Week 50.
- W50-Infliximab + Placebo: Placebo (PBO) oral capsules daily and Infliximab (IFX) infusions 5 mg/kg Week 30 through Week 50.
- W50-Infliximab + Azathioprine: Azathioprine (AZA) oral capsules daily 2.5 mg/kg/day and Infliximab (IFX) infusions 5 mg/kg Week 30 through Week 50.
- OLE-Azathioprine + Placebo/Infliximab: Azathioprine (AZA) oral capsules daily 2.5mg/kg/day and Placebo (PBO) infusion through Week 50. Infliximab (IFX) infusions 5mg/kg in one year country specific (UE and Israel) Open-Label Extension.
- OLE-Infliximab + Placebo/Infliximab: Placebo (PBO) oral capsules daily and infliximab (IFX) infusions 5mg/kg through Week 50. Infliximab (IFX) infusions 5mg/kg in one year country specific (UE and Israel) Open-Label Extension.
- OLE-Infliximab + Azathioprine/Infliximab: Azathioprine (AZA) oral capsules daily 2.5mg/kg/day and infliximab (IFX) infusions 5mg/kg through Week 50. Infliximab (IFX) infusions 5mg/kg in one year country specific (UE and Israel) Open-Label Extension.
Arm/Group | W30-Azathioprine + Placebo | W30-Infliximab + Placebo | W30-Infliximab + Azathioprine | W50-Azathioprine + Placebo | W50-Infliximab + Placebo | W50-Infliximab + Azathioprine | OLE-Azathioprine + Placebo/Infliximab | OLE-Infliximab + Placebo/Infliximab | OLE-Infliximab + Azathioprine/Infliximab
Serious Adverse Events (participants affected / at risk) | 39/161 | 26/163 | 25/179 | 5/75 | 15/97 | 2/108 | 1/8 | 1/18 | 3/17
Other Adverse Events (participants affected / at risk) | 120/161 | 122/163 | 133/179 | 44/75 | 69/97 | 61/108 | 7/8 | 16/18 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | W30-Azathioprine + Placebo (N=161) | W30-Infliximab + Placebo (N=163) | W30-Infliximab + Azathioprine (N=179) | W50-Azathioprine + Placebo (N=75) | W50-Infliximab + Placebo (N=97) | W50-Infliximab + Azathioprine (N=108) | OLE-Azathioprine + Placebo/Infliximab (N=8) | OLE-Infliximab + Placebo/Infliximab (N=18) | OLE-Infliximab + Azathioprine/Infliximab (N=17)
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Papilloedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 4 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal Fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colonic Stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Crohn's Disease (Gastrointestinal disorders) | 12 | 7 | 6 | 1 | 9 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal Stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolonic Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileal Stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal Fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal Stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 4 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Small Intestinal Stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis Acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactoid Reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Abscess (Infections and infestations) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abscess Intestinal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Campylobacter Intestinal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perirectal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia Legionella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomembranous Colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psoas Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retroperitoneal Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anastomotic Leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crush Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine with Aura (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conversion Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urethral Stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Miscarriage of Partner (Social circumstances) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | W30-Azathioprine + Placebo (N=161) | W30-Infliximab + Placebo (N=163) | W30-Infliximab + Azathioprine (N=179) | W50-Azathioprine + Placebo (N=75) | W50-Infliximab + Placebo (N=97) | W50-Infliximab + Azathioprine (N=108) | OLE-Azathioprine + Placebo/Infliximab (N=8) | OLE-Infliximab + Placebo/Infliximab (N=18) | OLE-Infliximab + Azathioprine/Infliximab (N=17)
Anaemia (Blood and lymphatic system disorders) | 5 | 4 | 2 | 1 | 2 | 1 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 10 | 1 | 0 | 2 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Amaurosis Fugax (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 1 | 1 | 0 | 1 | 4 | 0 | 0 | 1
Eyelids Pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular Hyperaemia (Eye disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Panophthalmitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uveitis (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 3 | 7 | 4 | 2 | 1 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 23 | 34 | 24 | 3 | 11 | 10 | 3 | 5 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 8 | 8 | 12 | 1 | 3 | 1 | 1 | 4 | 2
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Anal Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphthous Stomatitis (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 5 | 5 | 0 | 2 | 1 | 0 | 2 | 1
Crohn's Disease (Gastrointestinal disorders) | 14 | 7 | 10 | 4 | 10 | 6 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 11 | 14 | 11 | 2 | 7 | 6 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 4 | 9 | 2 | 1 | 1 | 0 | 1 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal Sounds Abnormal (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 2 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 46 | 27 | 39 | 7 | 11 | 6 | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 24 | 13 | 14 | 5 | 11 | 1 | 0 | 1 | 0
Chest Discomfort (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cyst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 22 | 21 | 24 | 5 | 4 | 4 | 2 | 4 | 6
Inflammation (General disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Influenza Like Illness (General disorders) | 2 | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 0
Malaise (General disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Oedema Peripheral (General disorders) | 3 | 3 | 4 | 2 | 0 | 4 | 0 | 0 | 1
Pyrexia (General disorders) | 16 | 10 | 13 | 1 | 6 | 5 | 1 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal Allergy (Immune system disorders) | 1 | 4 | 0 | 0 | 2 | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 2 | 2 | 8 | 4 | 1 | 0 | 1 | 0 | 1
Ear Infection (Infections and infestations) | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Fungal Infection (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 3 | 2 | 4 | 2 | 0 | 3 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 7 | 3 | 2 | 1 | 3 | 1 | 1 | 2 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Impetigo (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 8 | 6 | 3 | 1 | 3 | 2 | 3 | 3
Laryngitis (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 15 | 13 | 16 | 11 | 6 | 9 | 4 | 3 | 3
Oral Herpes (Infections and infestations) | 3 | 4 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 8 | 2 | 0 | 2 | 2 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 4 | 2 | 4 | 1 | 1 | 0 | 1 | 1 | 1
Sinusitis (Infections and infestations) | 5 | 2 | 6 | 3 | 6 | 1 | 1 | 1 | 1
Tinea Pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Tooth Abscess (Infections and infestations) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 3 | 9 | 4 | 4 | 1 | 0 | 0 | 1
Vulvovaginal Mycotic Infection (Infections and infestations) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Face Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 3 | 8 | 6 | 0 | 0 | 2 | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 2 | 6 | 6 | 1 | 0 | 1 | 0 | 0 | 1
Blood Albumin Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
C-Reactive Protein Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
C-Reactive Protein Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic Enzyme Increased (Investigations) | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Liver Function Test Abnormal (Investigations) | 3 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Weight Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 23 | 17 | 7 | 10 | 5 | 3 | 5 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 6 | 5 | 2 | 5 | 4 | 2 | 0 | 1
Lupus-Like Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 8 | 2 | 0 | 2 | 0 | 0 | 2 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 | 1 | 0 | 2 | 0 | 0 | 1
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign Neoplasm of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 11 | 10 | 1 | 2 | 0 | 1 | 2 | 0
Headache (Nervous system disorders) | 19 | 22 | 22 | 4 | 9 | 4 | 2 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 4 | 0 | 0 | 2 | 1 | 0 | 2 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Syncope Vasovagal (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 3 | 2 | 0 | 1 | 1 | 0 | 1 | 0
Depressed Mood (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 4 | 5 | 1 | 0 | 2 | 2 | 0 | 1 | 1
Fear (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 5 | 4 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Sleep Disorder (Psychiatric disorders) | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 4 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 11 | 2 | 4 | 1 | 3 | 0 | 3 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5 | 1 | 1 | 1 | 0 | 1 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 12 | 5 | 1 | 2 | 3 | 2 | 1 | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 3 | 3 | 4 | 0 | 0 | 3 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 7 | 7 | 1 | 0 | 1 | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 1 | 3 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 4 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Pain of Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Pityriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 2 | 3 | 1 | 1 | 0 | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 9 | 7 | 9 | 0 | 1 | 2 | 1 | 1 | 0
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pregnancy of Partner (Social circumstances) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Tooth Extraction (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 3 | 5 | 3 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days